CLINICAL TRIAL: NCT02187003
Title: A Phase 3, Multicenter ,Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Rivipansel (GMI-1070) in the Treatment of Vaso-Occlusive Crisis in Hospitalized Subjects With Sickle Cell Disease
Brief Title: Efficacy and Safety of Rivipansel (GMI-1070) in the Treatment of Vaso-Occlusive Crisis in Hospitalized Subjects With Sickle Cell Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biossil Inc. (Industry)
Collaborators: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B5201002; RESET (Other: Alias Study Number)
Record Dates: First submitted 2014-06-12; First posted 2014-07-10 (Estimated); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Disorders; pain crisis; vaso-occlusive crisis; rivipansel; GMI-1070; selectin inhibitor; SCD; VOC
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — rivipansel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rivipansel Treatment Arm (Experimental)
  Interventions: Drug: Rivipansel
- Placebo Treatment Arm (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rivipansel — Rivipansel (GMI-1070) will be infused intravenously every 12 hours up to 15 doses maximum. Subjects aged 12 and over who weigh more than 40 kilograms will receive a dose of 1680 mg of rivipansel, followed by a dose of 840 mg of rivipansel every 12 hours. All subjects aged 6 to 11 years and any subject who weighs 40 kilograms or less, will receive weight-based dosing (mg/kg) of 40 mg/kg of rivipansel (maximum of 1680 mg) followed by a dose of 20 mg/kg of rivipansel (maximum of 840 mg) every 12 hours.
  Other Names: GMI-1070
  Arms: Rivipansel Treatment Arm
Other: Placebo — Placebo (phosphate buffered saline) will be infused intravenously every 12 hours up to 15 doses maximum.
  Other Names: phosphate buffered saline (PBS)
  Arms: Placebo Treatment Arm

SUMMARY:
This is a clinical study evaluating the efficacy and safety of rivipansel (GMI-1070) in treating subjects with sickle cell disease (SCD) who are 6 years of age or older experiencing a pain crisis necessitating hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 years of age.
* Documented diagnosis of sickle cell disease.
* Diagnosis of vaso-occlusive crisis necessitating admission to the hospital with treatment including IV opioids.
* Able to receive the first dose of study drug within 24 hours from the administration of IV opioids.

Exclusion Criteria:

* Serious systemic infection
* Acute Chest Syndrome
* Serious concomitant medical problems (for example, stroke)
* SCD pain atypical of VOC
* Severe renal or hepatic impairment
* Chronic pain rather than a presentation of acute VOC

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (138):
- United States (123):
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - Arkansas Children's Hospital Research Pharmacy, Little Rock, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UC Davis Medical Center Main Hospital, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado CTRC, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Howard University Center for Sickle Cell Disease, Washington D.C., District of Columbia
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Davis Cancer Pavillion and Shands Med Plaza, Gainesville, Florida
  - UF Health Shands Cancer Hospital, Gainesville, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University Of Miami, Miami, Florida
  - Investigational Drug Service Tampa General Hospital, Tampa, Florida
  - Tampa General Hospital Center of Research Excellence, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Children's Hematology and Oncology Associates, West Palm Beach, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta Aflac Cancer and Blood Disorders Center, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia
  - Children's Healthcare of Atlanta: Scottish Rite Campus, Atlanta, Georgia
  - Augusta University Clinical Research Pharmacy, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Augusta University, Augusta, Georgia
  - Memorial Family Medicine Ctr. @Memorial Health Univ Med Ct, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - The University of Chicago/Comer Children's Hospital, Chicago, Illinois
  - University of Chicago, Investigational Drug Service Pharmacy, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Norton Children´s Hospital, Louisville, Kentucky
  - The Novak Center for Children's Health, Louisville, Kentucky
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - University of Louisville Physicians Pediatric Hematology Oncology, Louisville, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - St. Jude Affiliate Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group-Medical Oncology, Baton Rouge, Louisiana
  - University of Maryland Medical System Investigational Pharmacy, Baltimore, Maryland
  - University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins Medicine, Baltimore, Maryland
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Center for Clinical Investigation, Brigham & Women's Hospital, Boston, Massachusetts
  - Investigational Drug Services, Boston, Massachusetts
  - Boston Medical Center E7E, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Detroit Medical Center Pharmacy, Detroit, Michigan
  - Wayne State University / Detroit Receiving Hospital, Detroit, Michigan
  - University of Mississippi Medical Center-Outpatient Clinical Research Unit, Jackson, Mississippi
  - University Of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Center for Outpatient Health, St Louis, Missouri
  - Barnes-Jewish Hospital Department of Pharmacy, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Bristol Myers Squibb Children's Hospital at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rutgers Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - Kings County Hospital Center - Pharmacy Department, Brooklyn, New York
  - Kings County Hospital Center, Brooklyn, New York
  - State University of New York (SUNY) - Downstate Medical Center, Brooklyn, New York
  - SUNY Downstate Medical Center University Hospital of Brooklyn, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center Research Pharmacy, New York, New York
  - MS CHONY Pediatric Emergency Department, New York, New York
  - MS CHONY Pediatric Hematology/Oncology Unit, New York, New York
  - Staten Island University Hospital, Staten Island, New York
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University Brody School of Medicine, Greenville, North Carolina
  - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - University of Cincinnati Medical Center/ Investigational Pharmacy, Cincinnati, Ohio
  - University of Cincinnati Medical Center/Research Office, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Cincinnati Physicians Company LLC, Cincinnati, Ohio
  - University of Cincinnati- Hoxworth Building, Cincinnati, Ohio
  - UC Health Ridgeway Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center East, Columbus, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - The Ohio State University Investigational Drug Services, Columbus, Ohio
  - The Ohio State University James Comprehensive Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Five Rivers Medical Surgical Health Center, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Rhode Island Hospital-Pharmacy Service, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina - Hospital, Charleston, South Carolina
  - Medical University of South Carolina Lifespan Comprehensive Sickle Cell Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Investigational Drug Services, Charleston, South Carolina
  - Cook Children's Hematology and Oncology Center, Fort Worth, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Cook Children's Hematology and Oncology Center-Grapevine, Grapevine, Texas
  - Texas Children's Hospital - Clinical Research Center, Houston, Texas
  - Texas Children´s Hospital, Houston, Texas
  - University of Texas Medical School, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Main Hospital - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Commonwealth University-Investigational Drug Services, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (15):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Miseracordia Community Hospital, Edmonton, Alberta
  - Kaye Edmonton Clinic 3 C, Edmonton, Alberta
  - University of Alberta Hospital, Pharmacy Services, Edmonton, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Research transition Facility, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Children's Hospital Of Eastern Ontario, Ottawa, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - McGill University Health Centre, Royal Victoria Hospital, Montreal, Quebec
  - The Montreal Children's Hospital/ McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dampier CD, Telen MJ, Wun T, Brown RC, Desai P, El Rassi F, Fuh B, Kanter J, Pastore Y, Rothman J, Taylor JG, Readett D, Sivamurthy KM, Tammara B, Tseng LJ, Lozier JN, Thackray H, Magnani JL, Hassell KL; RESET Investigators. A randomized clinical trial of the efficacy and safety of rivipansel for sickle cell vaso-occlusive crisis. Blood. 2023 Jan 12;141(2):168-179. doi: 10.1182/blood.2022015797. PMID 35981565
- [Derived] Rebelo AL, Chevalier MT, Russo L, Pandit A. Role and therapeutic implications of protein glycosylation in neuroinflammation. Trends Mol Med. 2022 Apr;28(4):270-289. doi: 10.1016/j.molmed.2022.01.004. Epub 2022 Feb 1. PMID 35120836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, blinded study to treat subjects >=6 years of age with SCD, experiencing an acute VOC event requiring hospitalization. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population in alignment with the primary study objective.
Pre-assignment Details: Due to the short duration of time allowed to dose upon a VOC event, an optional screening may have occurred while the participant was well. Patients were neither enrolled nor randomized to study treatment until a VOC occurred, at which time the formal assessment of eligibility for enrollment into the study was performed. Of the 475 screened participants, 345 participants experiencing an acute VOC event were randomized.
Groups:
- Rivipansel Treatment Arm: Participants with sickle cell disease (SCD) received intravenous (IV) infusion of rivipansel while hospitalized for treatment of a vaso-occlusive crisis (VOC). Participants aged >=12 years, with body weight >40 kilogram (kg) received a loading dose of 1680 milligram (mg) rivipansel on Day 1 followed by maintenance doses of 840 mg rivipansel administered at 12 hourly intervals.
  Participants aged 6 to 11 years or any participant weighing <=40 kg received a loading dose of 40 milligram per kilogram body weight (mg/kg) rivipansel on Day 1 (maximum of 1680 mg) followed by maintenance doses of 20 mg/kg rivipansel (maximum of 840 mg) administered at 12 hourly intervals. Participants received rivipansel until they met the protocol-defined criteria for readiness-for-discharge from hospital or up to a maximum of 15 doses (1 loading dose and 14 maintenance doses), whichever occurred first. Dosing therefore continued for a maximum of 8 days.
- Placebo Treatment Arm: Participants with SCD received IV infusion of placebo (matched to rivipansel infusion) while hospitalized for treatment of a VOC. Participants received placebo on the same schedule used for rivipansel until they met the protocol-defined criteria for readiness-for- discharge from hospital or up to a maximum of 15 doses (1 loading dose and 14 maintenance doses), whichever occurred first. Dosing therefore continued for a maximum of 8 days
Period: Overall Study
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Started | 173 | 172
Treated | 162 | 158
Completed | 146 | 141
Not Completed | 27 | 31
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 14 | 10
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Protocol Violation | 2 | 4
Not completed — Other | 5 | 5
Not completed — Withdrawal by Parent/Guardian | 1 | 5

BASELINE CHARACTERISTICS:
Population: Full analysis set population included all participants who were randomized in the study. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population in alignment with the primary study objective.
  Full analysis set population included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm | Total
Number analyzed (Participants) | 173 | 172 | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.00 (10.61) | 21.34 (10.20) | 21.67 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 99 | 183
  Male | 89 | 73 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 16 | 23
  Not Hispanic or Latino | 165 | 155 | 320
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 167 | 159 | 326
  Race: White | 0 | 6 | 6
  Race: Other | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Time to Readiness for Discharge From Hospital
Description: Time to readiness-for-discharge from hospital was defined as the difference (in hours) between the time and date when all criteria for readiness-for-discharge were met and the start time and date of the first infusion (loading dose) of study drug. Criteria for readiness-for-discharge were met when all of the applicable 6 criteria (in relation to treatment of VOC and complications related to the VOC) were documented to have occurred. The six criteria were: 1) only oral pain medication was required, 2) acute complications related to the VOC (such as acute chest syndrome, stroke, priapism) had resolved to the extent that management could be in an outpatient setting, 3) IV opioids had been discontinued, 4) IV hydration had been discontinued, 5) IV antibiotics had been discontinued and 6) red blood cell (RBC) transfusion was no longer required for treatment of this VOC.
Time Frame: Day 1 up to the latest day when all 6 criteria of readiness-for-discharge were met (up to an average of Day 8)
Population: Full analysis set population included all participants who were randomized in the study. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population in alignment with the primary study objective.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 173 | 172
Hours | 87.78 [65.68 to 100.15] | 93.47 [74.67 to 109.73]
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; A Cox proportional hazards regression model with age group and genotype group as stratification covariates was used to estimate the hazard ratio (Placebo/Rivipansel) and the corresponding 95 percent (%) confidence interval (CI). A stratified log-rank test with age group and genotype group as stratification variables was performed to evaluate P value; Test type: Superiority; p = 0.7944, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.22]

2. Secondary Outcome: Time to Discharge From Hospital
Description: Time to discharge from hospital was defined as the difference (in hours) between the time and date of the hospital discharge order from a qualified healthcare provider and the start time and date of the first infusion (loading dose) of study drug.
Time Frame: Day 1 up to the latest day when the order of hospital discharge was issued by a qualified healthcare provider (up to an average of Day 8)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 173 | 172
Hours | 86.75 [71.25 to 98.72] | 90.67 [72.10 to 108.62]
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; A Cox proportional hazards regression model with age group and genotype group as stratification covariates was used to estimate the hazard ratio (Placebo/Rivipansel) and the corresponding 95% CI. A stratified log-rank test with age group and genotype group as stratification variables was performed to evaluate P- value; Test type: Superiority; p = 0.7156, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.77 to 1.19]

3. Secondary Outcome: Cumulative Intravenous (IV) Opioids Consumption From Time of Loading Dose of Study Drug to Discharge From Hospital
Description: Cumulative IV opioid consumption was reported as cumulative IV opioid use (standardized using morphine equivalent units [MEU]), from the start of the first infusion (loading dose) of study drug until hospital discharge.
Time Frame: Day 1 up to the latest day when IV opioid was discontinued (up to an average of Day 8)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: MEU per kg
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 173 | 172
MEU per kg | 2.30 [0.68 to 6.03] | 2.36 [0.55 to 6.99]
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; The difference in medians (Rivipansel- Placebo) was estimated by the difference of treatment medians from summary statistics. The corresponding 95% CI was estimated by a bootstrap method with stratification for age and genotype groups. P-value was from analysis of covariance (ANCOVA) model based on rank-transformed values using age group and genotype group as the stratification covariates; Test type: Superiority; p = 0.8520, ANCOVA; Mean Difference (Net) = -0.06, 95% CI 2-sided [-1.27 to 0.88]

4. Secondary Outcome: Time to Discontinuation of Intravenous (IV) Opioids
Description: Time to discontinuation of IV opioids was defined as the difference (in hours) between the stop time and date of the latest IV opioid dose and the start time and date of the first infusion (loading dose) of study drug.
Time Frame: Day 1 up to the latest day when IV opioid was discontinued (up to an average of Day 8)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 173 | 172
Hours | 67.20 [53.32 to 80.53] | 68.45 [53.75 to 84.97]
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.8593, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.82 to 1.26]

5. Secondary Outcome: Cumulative Intravenous (IV) Opioids Consumption Within First 24 Hours Post-Loading Dose of Study Drug
Description: Cumulative IV opioid consumption (standardized using MEU) was reported as IV opioid use in the first 24 hours from the start time of the first IV infusion (loading dose) of study drug.
Time Frame: 24 hours post first IV infusion of loading dose of study drug on Day 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: MEU per kg
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 173 | 172
MEU per kg | 0.80 [0.37 to 1.39] | 0.82 [0.40 to 1.56]
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; The difference in medians (Rivipansel- Placebo) was estimated by the difference of treatment medians from summary statistics. The corresponding 95% CI was estimated by a bootstrap method with stratification for age and genotype groups. P value was from ANCOVA model based on rank-transformed values using age group and genotype group as the stratification covariates; Test type: Superiority; p = 0.9332, ANCOVA; Median Difference (Final Values) = -0.02, 95% CI 2-sided [-0.13 to 0.16]

6. Secondary Outcome: Percentage of Participants Re-hospitalized for Vaso-Occlusive Crisis (VOC) Within 3 Days of Discharge From Hospital
Description: Percentage of participants who were re-hospitalized for a vaso-occlusive crisis (VOC) within 3 days of discharge from hospital are reported.
Time Frame: Within 3 days of discharge from hospital, where discharge from hospital was any day from Day 1 to an average of Day 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 173 | 172
Participants | 3 | 5
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; P values and 95% CI for the difference in percentages were based on the exact method by Chan and Zhang; Test type: Superiority; p = 0.5349, Chan and Zhang; Difference in percentage of participants = -1.17, 95% CI 2-sided [-5.19 to 2.46]

7. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) as Per Genotype
Description: AE: any untoward medical occurrence in a participant who received investigational product without regard to possibility of a causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. An adverse event was considered a treatment-emergent adverse event (TEAE) if the event started during the effective duration of treatment (all events that started on or after the first dosing). AEs included both serious and non-serious adverse events.
  Participants with AEs and SAEs were categorized by genotype categories. Category 1= participants with hemoglobin SS, hemoglobin S beta0 thalassemia and hemoglobin SD; category 2= participants with hemoglobin SC, hemoglobin S beta+ thalassemia and hemoglobin S-Variant (other than HbSD).
Time Frame: Day 1 up to the 35-day post discharge visit (up to an average of Day 43)
Population: Safety analysis set population included all participants who received at least 1 infusion of study drug. Here, "Number Analyzed" signifies number of participants evaluable for specified rows. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Participants
  Treatment Emergent AEs: number analyzed (Participants) | 143 | 130
  Treatment Emergent AEs: Genotype Category 1 | 112 | 101
  Treatment Emergent AEs: Genotype Category 2 | 31 | 29
  Treatment Emergent SAEs: number analyzed (Participants) | 52 | 49
  Treatment Emergent SAEs: Genotype Category 1 | 44 | 40
  Treatment Emergent SAEs: Genotype Category 2 | 8 | 9

8. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Event (AEs) as Per Severity
Description: AE: any untoward medical occurrence in a participant who received investigational product without regard to possibility of a causal relationship. AEs were classified according to the severity in 3 categories a) mild - AEs did not interfere with participant's usual function, b) moderate - AEs interfered to some extent with participant's usual function, c) severe - AEs interfered significantly with participant's usual function.
Time Frame: Day 1 up to the 35-day post discharge visit (up to an average of Day 43)
Population: Safety analysis set population included all participants who received at least 1 infusion of study drug. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Participants
  Mild | 49 | 43
  Moderate | 58 | 53
  Severe | 36 | 34

9. Other Pre Specified Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Hematology: hemoglobin, hematocrit, erythrocytes <0.8*lower limit of normal (LLN), reticulocytes <0.5*LLN >1.5*ULN, platelets<0.5*LLN>1.75*upper limit of normal (ULN), reticulocytes/erythrocytes<0.5*LLN>1.5*ULN, leukocytes <0.6*LLN >1.5*ULN, lymphocytes, lymphocytes/leukocytes, neutrophils, neutrophils/leukocytes <0.8*LLN >1.2*ULN, basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes, monocytes monocytes/leukocytes >1.2*ULN. Clinical chemistry: bilirubin, direct, bilirubin, indirect bilirubin>1.5*ULN, aspartate aminotransferase (AT), alanine AT, lactate dehydrogenase, alkaline phosphatase>3.0*ULN, urea nitrogen, urea, creatinine >1.3*ULN, sodium<0.95*LLN>1.05*ULN, potassium, chloride, bicarbonate<0.9*LLN>1.1*ULN, glucose<0.6*LLN>1.5*ULN, estimated glomerular filtration rate <=60. Urinalysis: urine glucose, ketones, urine protein, urine hemoglobin, nitrite, leukocyte esterase >=1.
Time Frame: Day 1 up to the 35-day post discharge visit (up to an average of Day 43)
Population: Safety analysis set population included all participants who received at least 1 infusion of study drug. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 161 | 154
Participants | 98 | 107

10. Other Pre Specified Outcome: Number of Participants With Increase in Grades From Baseline in Clinical Laboratory Parameters Over the Study
Description: Hemoglobin(grade [G] 0:>11g/dl,G1:>9-11g/dl,G2:>7-9g/dl,G3:5-7g/dl,G4:<5g/dl),reticulocytes count(G0:<1%,G1:1-5%,G2:>5-10%,G3:>10-20%,G4:>20%),leukocytes(G0:<=upper limit of normal [ULN],G1:>ULN-15,000/mm^3,G2:>15,000- 20,000/mm^3,G3:>20,000- 50,000/mm^, G4:>50,000/mm^3),neutrophils(G0:>=LLN, G1:<LLN-1,500/mm^3, G2:<1,500-1,000/mm^3, G3:<1,000-500/mm^3, G4:<500/mm^3),blood urea nitrogen, creatinine(G0:<=ULN, G1:>ULN-1.5*UL, G2:>1.5-3.0*ULN, G3:>3.0*ULN, G4:>6.0*ULN), lactate dehydrogenase, alanine transaminase, aspartate aminotransferase(G0:<=ULN, G1:>ULN-3.0*ULN, G2:>3.0-5.0*ULN, G3:>5.0-20.0*ULN, G4:>20.0*ULN), bilirubin(G0:<=ULN, G1:>ULN-1.5*ULN, G2:>1.5-3.0*ULN, G3:>3.0-10.0*ULN, G4:>10.0*ULN), urine protein(G0:0-15mg/dL, G1:>15-30mg/dL, G2:>30-100mg/dL, G3:>100-300mg/dL, G4:>300mg/dL), platelet(G0:>=150K, G1:>=100K-<150K, G2:>=50K <100K, G3:<50K), eGFR (G0:>=90 mL/min/1.73m^2, G1:>=60-<90mL/min/1.73m^2, G2:>=30-<60mL/min/1.73m^2, G3:>=15-<30mL/min/1.73m^2, G4:<15 mL/min/1.73m^2)
Time Frame: Baseline up to the 35-day post discharge visit (up to an average of Day 43)
Population: Safety analysis set population included all participants who received at least 1 infusion of drug. Overall Number of Participants Analyzed signifies participants evaluable for this outcome measure; Number Analyzed signifies participants evaluable for specific rows. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population.
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 161 | 154
Participants
  Hemoglobin : >=1 grade: number analyzed (Participants) | 153 | 145
  Hemoglobin : >=1 grade | 60 | 47
  Hemoglobin : >=2 grade: number analyzed (Participants) | 153 | 145
  Hemoglobin : >=2 grade | 3 | 5
  Hemoglobin : >=3 grade: number analyzed (Participants) | 153 | 145
  Hemoglobin : >=3 grade | 0 | 0
  Hemoglobin : >=4 grade: number analyzed (Participants) | 153 | 145
  Hemoglobin : >=4 grade | 0 | 0
  Reticulocytes/Erythrocytes : >=1 grade: number analyzed (Participants) | 81 | 82
  Reticulocytes/Erythrocytes : >=1 grade | 12 | 9
  Reticulocytes/Erythrocytes : >=2 grade: number analyzed (Participants) | 81 | 82
  Reticulocytes/Erythrocytes : >=2 grade | 1 | 2
  Reticulocytes/Erythrocytes : >=3 grade: number analyzed (Participants) | 81 | 82
  Reticulocytes/Erythrocytes : >=3 grade | 1 | 0
  Reticulocytes/Erythrocytes : >=4 grade: number analyzed (Participants) | 81 | 82
  Reticulocytes/Erythrocytes : >=4 grade | 0 | 0
  Platelets : >=1 grade: number analyzed (Participants) | 154 | 145
  Platelets : >=1 grade | 11 | 7
  Platelets : >=2 grade: number analyzed (Participants) | 154 | 145
  Platelets : >=2 grade | 1 | 1
  Platelets : >=3 grade: number analyzed (Participants) | 154 | 145
  Platelets : >=3 grade | 0 | 0
  Platelets : >=4 grade: number analyzed (Participants) | 154 | 145
  Platelets : >=4 grade | 0 | 0
  Leukocytes : >=1 grade: number analyzed (Participants) | 153 | 145
  Leukocytes : >=1 grade | 20 | 16
  Leukocytes : >=2 grade: number analyzed (Participants) | 153 | 145
  Leukocytes : >=2 grade | 4 | 3
  Leukocytes : >=3 grade: number analyzed (Participants) | 153 | 145
  Leukocytes : >=3 grade | 1 | 0
  Leukocytes : >=4 grade: number analyzed (Participants) | 153 | 145
  Leukocytes : >=4 grade | 0 | 0
  Direct Bilirubin : >=1 grade: number analyzed (Participants) | 121 | 124
  Direct Bilirubin : >=1 grade | 32 | 28
  Direct Bilirubin : >=2 grade: number analyzed (Participants) | 121 | 124
  Direct Bilirubin : >=2 grade | 7 | 10
  Direct Bilirubin : >=3 grade: number analyzed (Participants) | 121 | 124
  Direct Bilirubin : >=3 grade | 1 | 1
  Direct Bilirubin : >=4 grade: number analyzed (Participants) | 121 | 124
  Direct Bilirubin : >=4 grade | 0 | 1
  Indirect Bilirubin : >=1 grade: number analyzed (Participants) | 118 | 123
  Indirect Bilirubin : >=1 grade | 23 | 20
  Indirect Bilirubin : >=2 grade: number analyzed (Participants) | 118 | 123
  Indirect Bilirubin : >=2 grade | 1 | 2
  Indirect Bilirubin : >=3 grade: number analyzed (Participants) | 118 | 123
  Indirect Bilirubin : >=3 grade | 0 | 0
  Indirect Bilirubin : >=4 grade: number analyzed (Participants) | 118 | 123
  Indirect Bilirubin : >=4 grade | 0 | 0
  Aspartate Aminotransferase : >=1 grade: number analyzed (Participants) | 140 | 140
  Aspartate Aminotransferase : >=1 grade | 22 | 25
  Aspartate Aminotransferase : >=2 grade: number analyzed (Participants) | 140 | 140
  Aspartate Aminotransferase : >=2 grade | 0 | 2
  Aspartate Aminotransferase : >=3 grade: number analyzed (Participants) | 140 | 140
  Aspartate Aminotransferase : >=3 grade | 0 | 0
  Aspartate Aminotransferase : >=4 grade: number analyzed (Participants) | 140 | 140
  Aspartate Aminotransferase : >=4 grade | 0 | 0
  Alanine Aminotransferase : >=1 grade: number analyzed (Participants) | 142 | 140
  Alanine Aminotransferase : >=1 grade | 23 | 19
  Alanine Aminotransferase : >=2 grade: number analyzed (Participants) | 142 | 140
  Alanine Aminotransferase : >=2 grade | 1 | 4
  Alanine Aminotransferase : >=3 grade: number analyzed (Participants) | 142 | 140
  Alanine Aminotransferase : >=3 grade | 0 | 0
  Alanine Aminotransferase : >=4 grade: number analyzed (Participants) | 142 | 140
  Alanine Aminotransferase : >=4 grade | 0 | 0
  Lactate Dehydrogenase : >=1 grade: number analyzed (Participants) | 134 | 125
  Lactate Dehydrogenase : >=1 grade | 16 | 15
  Lactate Dehydrogenase : >=2 grade: number analyzed (Participants) | 134 | 125
  Lactate Dehydrogenase : >=2 grade | 0 | 1
  Lactate Dehydrogenase : >=3 grade: number analyzed (Participants) | 134 | 125
  Lactate Dehydrogenase : >=3 grade | 0 | 0
  Lactate Dehydrogenase : >=4 grade: number analyzed (Participants) | 134 | 125
  Lactate Dehydrogenase : >=4 grade | 0 | 0
  Urea Nitrogen : >=1 grade: number analyzed (Participants) | 139 | 132
  Urea Nitrogen : >=1 grade | 2 | 1
  Urea Nitrogen : >=2 grade: number analyzed (Participants) | 139 | 132
  Urea Nitrogen : >=2 grade | 0 | 0
  Urea Nitrogen : >=3 grade: number analyzed (Participants) | 139 | 132
  Urea Nitrogen : >=3 grade | 0 | 0
  Urea Nitrogen : >=4 grade: number analyzed (Participants) | 139 | 132
  Urea Nitrogen : >=4 grade | 0 | 0
  Creatinine : >=1 grade: number analyzed (Participants) | 153 | 144
  Creatinine : >=1 grade | 0 | 1
  Creatinine : >=2 grade: number analyzed (Participants) | 153 | 144
  Creatinine : >=2 grade | 0 | 1
  Creatinine : >=3 grade: number analyzed (Participants) | 153 | 144
  Creatinine : >=3 grade | 0 | 0
  Creatinine : >=4 grade: number analyzed (Participants) | 153 | 144
  Creatinine : >=4 grade | 0 | 0
  Urine Protein : >=1 grade: number analyzed (Participants) | 109 | 99
  Urine Protein : >=1 grade | 3 | 0
  Urine Protein : >=2 grade: number analyzed (Participants) | 109 | 99
  Urine Protein : >=2 grade | 2 | 0
  Urine Protein : >=3 grade: number analyzed (Participants) | 109 | 99
  Urine Protein : >=3 grade | 0 | 0
  Urine Protein : >=4 grade: number analyzed (Participants) | 109 | 99
  Urine Protein : >=4 grade | 0 | 0
  Neutrophils : >=1 grade: number analyzed (Participants) | 96 | 94
  Neutrophils : >=1 grade | 3 | 2
  Neutrophils : >=2 grade: number analyzed (Participants) | 96 | 94
  Neutrophils : >=2 grade | 3 | 1
  Neutrophils : >=3 grade: number analyzed (Participants) | 96 | 94
  Neutrophils : >=3 grade | 0 | 1
  Neutrophils : >=4 grade: number analyzed (Participants) | 96 | 94
  Neutrophils : >=4 grade | 0 | 0
  eGFR : >=1 grade: number analyzed (Participants) | 153 | 144
  eGFR : >=1 grade | 4 | 6
  eGFR : >=2 grade: number analyzed (Participants) | 153 | 144
  eGFR : >=2 grade | 0 | 1
  eGFR : >=3 grade: number analyzed (Participants) | 153 | 144
  eGFR : >=3 grade | 0 | 0
  eGFR : >=4 grade: number analyzed (Participants) | 153 | 144
  eGFR : >=4 grade | 0 | 0

11. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Physical Examination
Description: Physical examination included assessment of the general appearance and the skin, head, ears, eyes, nose, mouth, throat, spine, neck, thyroid, chest, extremities, lymph nodes and abdomen (including liver and kidneys) plus the respiratory, cardiovascular, musculoskeletal, neurological and genitourinary systems. Clinical significance was assessed by the Investigator.
Time Frame: From Post-screening up to end of treatment (up to an average of Day 8), From Post-discharge up to 35 days post-discharge (up to an average of Day 43)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Participants
  Post-screening up to end of treatment: number analyzed (Participants) | 157 | 156
  Post-screening up to end of treatment | 38 | 41
  Post-discharge to 35 days post-discharge: number analyzed (Participants) | 160 | 155
  Post-discharge to 35 days post-discharge | 25 | 25

12. Other Pre Specified Outcome: Number of Participants With Treatment Related Changes From Baseline in Vital Signs Over the Study
Description: Vital signs included temperature, respiratory rate, pulse rate and systolic and diastolic blood pressure. Relatedness to treatment was assessed by the Investigator.
Time Frame: Baseline (Day 1) up to the 35-day post discharge visit (up to an average of Day 43)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Participants | 0 | 0

13. Other Pre Specified Outcome: Percentage of Participants With Adjudicated Acute Chest Syndrome (ACS)
Description: Investigator reported events of Acute Chest Syndrome (ACS) and other reported respiratory events were sent for adjudication by the Acute Chest Syndrome Safety Endpoint Adjudication Committee. The committee, which consisted of physicians with relevant SCD expertise, evaluated these events and determined whether they were consistent with cases of ACS.
Time Frame: Day 1 up to the 35-day post discharge visit (up to an average of Day 43)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Percentage of participants | 6.8 | 10.1
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; Test type: Superiority; p = 0.3020, Chan and Zhang; Risk Difference (RD) = -3.336, 95% CI 2-sided [-10.024 to 2.968]

14. Other Pre Specified Outcome: Percentage of Participants With Severe Adjudicated and/or Generalized Cutaneous Manifestations
Description: Investigator reported cutaneous events were sent for adjudication by the Cutaneous Manifestations Safety Endpoint Adjudication Committee. The committee, which consisted of dermatologists, evaluated these events and determined whether they were cases of severe and/or generalized cutaneous manifestations and specifically whether any event was consistent with Acute Generalized Exanthematous Pustulosis.
Time Frame: Day 1 up to the 35-day post discharge visit (up to an average of Day 43)
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Percentage of participants | 2.5 | 1.3
Statistical Analysis 1: Comparison: Rivipansel Treatment Arm vs Placebo Treatment Arm; Test type: Superiority; p = 0.5429, Chan and Zhang; Risk Difference (RD) = 1.203, 95% CI 2-sided [-2.379 to 5.104]

15. Other Pre Specified Outcome: Percentage of Participants Re-hospitalized for Vaso-Occlusive Crisis (VOC) Within 7, 14 and 30 Days of Discharge From Hospital
Description: Percentage of participants re-hospitalized for VOC within 7, 14 and 30 days of hospital discharge.
Time Frame: Within 7 days of discharge; Within 14 days of discharge; Within 30 days of discharge, where discharge from hospital was any day from Day 1 to an average of Day 8
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 162 | 158
Percentage of participants
  Within 7 Days | 3.7 | 5.7
  Within 14 Days | 6.8 | 8.9
  Within 30 Days | 16.0 | 17.1

ADVERSE EVENTS:
Time Frame: Day 1 up to the 35-day post discharge visit (up to an average of Day 43)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Safety analysis set population included all participants who received at least one 1 infusion of study drug. Participants aged 12 years and above were identified as Cohort 1 and participants aged 6-11 years were identified as Cohort 2; however, the primary analysis and study conclusions were based on the full study population.
Arm/Group | Rivipansel Treatment Arm | Placebo Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/158
Serious Adverse Events (participants affected / at risk) | 52/162 | 49/158
Other Adverse Events (participants affected / at risk) | 137/162 | 124/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivipansel Treatment Arm (N=162) | Placebo Treatment Arm (N=158)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 37 | 34
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 1 | 0
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Blood culture positive (Investigations) | 0 | 1
Chest X-ray abnormal (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivipansel Treatment Arm (N=162) | Placebo Treatment Arm (N=158)
Anaemia (Blood and lymphatic system disorders) | 18 | 11
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 12 | 17
Sickle cell disease (Congenital, familial and genetic disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Constipation (Gastrointestinal disorders) | 29 | 21
Diarrhoea (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 26 | 27
Vomiting (Gastrointestinal disorders) | 17 | 16
Chest pain (General disorders) | 9 | 8
Infusion site extravasation (General disorders) | 4 | 1
Oedema peripheral (General disorders) | 2 | 4
Pain (General disorders) | 6 | 6
Peripheral swelling (General disorders) | 3 | 4
Pyrexia (General disorders) | 29 | 33
Ocular icterus (Hepatobiliary disorders) | 3 | 4
Pneumonia (Infections and infestations) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Alanine aminotransferase increased (Investigations) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 6
Haematocrit decreased (Investigations) | 0 | 5
Haemoglobin decreased (Investigations) | 9 | 12
Oxygen saturation decreased (Investigations) | 8 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 8
Dizziness (Nervous system disorders) | 9 | 4
Headache (Nervous system disorders) | 18 | 29
Somnolence (Nervous system disorders) | 4 | 2
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 24 | 17
Rash (Skin and subcutaneous tissue disorders) | 8 | 6
Hypertension (Vascular disorders) | 5 | 0
Hypotension (Vascular disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT02187003/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT02187003/SAP_001.pdf